CLINICAL TRIAL: NCT03586310
Title: Evaluation of the Ear-EEG System for Sleep Monitoring in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Uneeg medical (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EarEEGSleep2018
Record Dates: First submitted 2018-03-16; First posted 2018-07-13 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2019-05

CONDITIONS: Sleep Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 nights with PSG (Other): For all subjects: 4 nights with polysomnography and ear-EEG
  Interventions: Device: ear-EEG
- 12 nights with ear-EEG (Other): For a subset of the subjects in arm the '4 nights with PSG', a second phase follows in which each subject sleeps 12 nights with only ear-EEG.
  If a night's recording is unsuccessful, for whatever reason, up to 6 additional nights may be attempted.
  Interventions: Device: ear-EEG

INTERVENTIONS:
Device: ear-EEG — soft silicone electrode array placed in each ear (outer ear-canal and concha), connected to a battery powered EEG amplifier.

SUMMARY:
Subjects sleep multiple nights in their own home, wearing actigraph, PSG (PolySomnoGraphy) and ear-EEG sensors. The object of the study is to determine the applicability of ear-EEG for sleep monitoring.

ELIGIBILITY:
Inclusion Criteria:

Informed consent obtained and letter of authority signed before any study related activities

Age 18-50 years

-

Exclusion Criteria:

1. BMI (body mass index) > 30
2. Previous stroke or cerebral haemorrhage and any other structural cerebral disease
3. Known or suspected abuse of alcohol or any other neuro-active substance
4. Use of hearing aid or cochlear implants
5. Allergic contact dermatitis caused by metals or generally prone to skin irritation
6. Narrow or malformed ear canals
7. Obstructive sleep apnea
8. History of sleep disorders or neurological diseases
9. Chronic pain
10. People judged incapable, by the investigator, of understanding the participant instruction or who are not capable of carrying through the investigation.
11. Use of medication known to influence the user's sleep (antidepressants, sedatives, antipsychotic-, and pain relieving medication)
12. Teeth grinding (bruxism)
13. Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Cohens kappa | At study completion (average of 6 months)
  The test outcome is a set of matched polysomnography and ear-EEG sleep measurements. From this will be generated an algorithm for automatic sleep scoring based on ear-EEG (using leave-one-subject-out cross validation). The primary outcome measure of the test is the correlation between the automatically generated hypnograms and those generated manually from the scalp recordings.
  The accuracy is quantified using Cohen's kappa, which is a number between -1 and 1. An average (across all recordings) above 0.4 would be a success for the test.
  As the training of the sleep scoring algorithm requires large amounts of data, it is necessary to use a large number of subjects (20) to estimate the viability of automatic sleep scoring from ear-EEG recordings. This also means that kappa values are calculated for all recordings at once when the measurements are done.
  This method for creating sleep scoring algorithms and quantifying their success is in line with standard procedure in this field.

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kidmose, Professor, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After publication of results, anonymized recordings will be made available to the scientific community.
Time Frame: We anticipate that data will be made available at some point in 2019.